CLINICAL TRIAL: NCT05628402
Title: Qualitative Study on Cognitive Mecanisms Involved in Exhibitionists's Acting Out
Brief Title: Exhibitionnists's Cognitive Mecanisms
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL22_0411
Record Dates: First submitted 2022-11-16; First posted 2022-11-28 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Paraphilic Disorders; Exhibitionism
Keywords: sex offender; sexual violence; acting out
MeSH Terms: conditions — Paraphilic Disorders; Exhibitionism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- exhibitionist patients
  Interventions: Other: Semi-structured interview

INTERVENTIONS:
Other: Semi-structured interview — The semi-structured interview will take place during a standard follow-up appointment with the therapist already treating the patient after the patient has agreed to participate in the study.

SUMMARY:
Exhibitionism is a paraphilia, which is defined according to the DSM 5. The estimated prevalence in men is between 2 to 4% (The prevalence of exhibitionistic disorder in females is even more uncertain but is generally believed to be much lower than in males).

At judiciary level: approximately 30% of apprehended male sex offenders are exhibitionists. They have the highest recidivism rate of any sex offender; about 20-50% are arrested again.

The studies are old and not very prolific on the subject of exhibition. The available data are lacking, there is no clinical evaluation scale for exhibitionism. The diagnosis is essentially based on facts with judicial characteristics "did patient show himself? ", "Does he enjoy showing off?". Investigators have no data on the cognitive distortions that support this particular acting out, the (specific) triggering factors and the potential psychological vulnerabilities of exhibitionists Some cognitive and sensory mechanisms may be involved in the origin and development of the processes underlying the act (Johnston and Ward 1996). The investigators will rely on the identification of anticipatory, relieving and permissive beliefs as a schema that can explain cognitive processes leading to acting out (Johnston and Ward, 1996). The goal is to apply this approach to exhibitionism. It should be noted that this model of thoughts (anticipatory, relieving and permissive) is taken up in the field of addiction. Exhibition is generally presented in the literature as a possible addictive disorder (Jon E. et al). The investigators will investigate whether there are specific factors precipitating exhibitionnism's acting out, other than the general precipitating factors or the recidivism risk factors known in sexual violence (SONAR, STATIC-99, PCL- R, SVR-20…). The investigators will also study the psychological vulnerabilies of these subjects.

ELIGIBILITY:
Inclusion Criteria:

* male > 18 years
* followed in Resource Centre for Interveners with Perpetrators of Sexual Violence of Montpellier UH
* exhibitionnists
* agree to participate

Exclusion Criteria:

* dementia
* severe intellectual desability
* decompensated psychiatric didease

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men followed for exhibitionism
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-09-06 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Self-questionnaire | Day 1 (inclusion)
  collective and personal representation on the phenomeon, self-reflexivity in relation to personality, self reflexivity in relation to body and sexuality, exploration of the lived expérience of exhbition, exploration of evolution in term of addiction

SECONDARY OUTCOMES:
Sexual Addiction Screening Test : SAST-Fr | Day 1
  The Sexual Addiction Screening Test (SAST) is designed to assist in the assessment of sexually compulsive or "addictive" behavior.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Montpellier : Lapeyronie CRIAVS, Montpellier, France

REFERENCES:
- [Result] Marais C, Song Y, Ferreira R, Aounti S, Duflos C, Baptista G, Pers YM. Evaluation of mindfulness based stress reduction in symptomatic knee or hip osteoarthritis patients: a pilot randomized controlled trial. BMC Rheumatol. 2022 May 30;6(1):46. doi: 10.1186/s41927-022-00277-9. PMID 35637515
- See also: open access — https://rdcu.be/cODwx